CLINICAL TRIAL: NCT06057142
Title: Fun Activities for Reciting Tang Poems to Promote Happiness in Primary School Ethnic Minority Students in Hong Kong
Brief Title: Reciting Tang Poems to Promote Happiness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Metropolitan University (Other)
Collaborators: Bestreben Drama Association Limited (Unknown)
Responsible Party: Principal Investigator, Dr Grace SUN Yuying, Assistant Professor, Hong Kong Metropolitan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HE-SF2023/21
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Acculturation; Happiness; Well-Being, Psychological; Ethnic Minority
Keywords: Tang poems; Happiness; Ethnic minority students
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This is a pilot pre-intervention trial without controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fun activities for reciting Tang poems (Experimental): The students will participate in three weekly sessions of Tang poem classes and one session of performance show. Each session lasts for 1.5 hours. Parents can sit in the class. A total of six poems will be taught by two experienced Chinese teachers.
  Interventions: Behavioral: Fun activities for reciting Tang poems

INTERVENTIONS:
Behavioral: Fun activities for reciting Tang poems — The students will participate in three weekly sessions of Tang poem classes and one session of performance show. Each session lasts for 1.5 hours. Parents can sit in the class. A total of six poems will be taught by two experienced Chinese teachers.

SUMMARY:
The ethnic minority population is increasing Hong Kong. Language learning is usually measured as one of the core indicators of acculturation. Chinese Tang poems use a specific mirror symmetry that could make people acquire unconscious learning. The goal of this pilot pre-post interventional trial with no controls is to explore the feasibility and preliminary evidence of the effectiveness of using fun activities for Tang poem reading to promote reciting and happiness in primary school ethnic minority and their families. Participants will be invited to participate in three Tang poetry recitation sessions and one participant performance session. The hypothesis is that participants with a greater number of successful recited poems will show higher happiness and enjoyment by students.

DETAILED DESCRIPTION:
Tang poems are not only for language learning but also induce people's positive emotions. Traditionally, some Chinese parents teach the very young kids to recite Tang poems even before the kids know how to read and write. Reciting Tang poems resembles singing a song without understanding the verses, and some kids can do so better than adults. Tang poems sound musical and should be easier to remember and recite than other texts. Learning and reciting poems at home could be happy and fun family activities in Chinese families. Whether using fun activities on small groups of kids in a community setting to promote Tang poem reciting and happiness could have the same effects of Tang poem reciting in Chinese kids is unknown for non-Chinese.

This is a pilot pre-post interventional trial with no controls, with 10 South Asian children in primary schools (Grades 1-2, age 6-9) being recruited in Phase I and 40-50 children in Phase II. In most primary schools, grades 1-2 students have not started learning Tang poems. Students and their parents will be actively approached by Hong Kong Christian Service (HKCS). An information sheet will be provided to the parents of eligible children, and their contact information will be asked. Parents give written consent if they agree for their children to participate. Parents will be invited to join the intervention sessions to show support for students' participation but they will only sit at the back of the room without active interaction and learning requirements.

The intervention comprises three 1.5-hour sessions of Tang poem reciting and one session for participant performances. Experienced instructors from Bestreben Drama Association Limited will lead each session, and adherence to the protocol will be assessed by independent reviewers. Participants will recite two poems per session, with adjustments based on performance. Body language, sound, images, and videos will be used, along with engaging games, to enhance motivation and memory. Participants will receive stamp/sticker collection books and be rewarded for their achievements. Parents are invited to attend the sessions to show support, their role will be passive, sitting at the back of the room without active interaction or learning requirements. A final session will include a 15-minute assessment of poem recitation skills, followed by a performance session where participants can recite any Tang poem. Family members are encouraged to participate, and awards will be granted to motivate and appreciate participants and their families.

In Phase I, assessments will include pre-session assessments (T0, T2, T4, and T6) and post-intervention assessments after each session (T1, T3, T5, and T7). A follow-up assessment (T8) will be conducted 12 weeks after the baseline to evaluate the sustainability of outcomes approximately one month after program completion. For the children in Phase II, assessments will only include T0, T5, T6, T7 and T8. Parents will complete questionnaires for themselves (Part II) and assisting their children (Part I). Parental presence and support will be acknowledged through supermarket coupon incentives.

The feasibility outcomes will be reported descriptively and narratively, including the recruitment rate, duration, and retention rate. Descriptive statistics, mean (standard deviation) for continuous outcomes, will be reported for the secondary outcomes. The investigators will use content analysis method to analyze the qualitative data from the in-depth interviews. It is expected that those fun activities for reciting Tang poems may help promoting happiness and enjoyment in primary school ethnic minority students in Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

* Ethnic minority children in primary schools (Grades 1-2, age 6-12)
* Able to communicate using either simple Cantonese or English
* With parental consent, and consent of the child as confirmed by the parent and our research team at the session

Exclusion Criteria:

* Physically or mentally unable to communicate
* Unwilling to participate regardless of parental consent
* Being involved in other similar activities or research
* Already proficient in Tang poems, being able to recite more than one poem

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2023-10-06 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Number of successful recited poems reported by independent observers. | T1: immediately after Session 1 (Week 1); T3: immediately after Session 2 (Week 2); T5: immediately after Session 3 (Week 3); T7: immediately after Session 4 (Week 7)
  Actual number of successful recited poems (over 80% wording are correct) assessed objectively by independent observers in session and on videos/photos.
Change in the number of successful recited poems reported subjectively by students. | T0: baseline; T2: right before Session 2 (Week 2); T4: right before Session 3 (Week 3); T6: right before Session 4 (Week 7); T8: Week 12
  Actual number of successful recited poems reported subjectively by students using a single-item question (How many Tang poems can you recite successfully (over 80% correct) at present).
Change in happiness reported subjectively by students. | T0: baseline; T2: right before Session 2 (Week 2); T4: right before Session 3 (Week 3); T6: right before Session 4 (Week 7); T8: Week 12
  Happiness reported subjectively by students (0 strongly disagree - 10 strongly agree) using a single-item question (I feel happy in general).
Change in happiness reported objectively by independent observers | T0: baseline; T2: right before Session 2 (Week 2); T4: right before Session 3 (Week 3); T6: right before Session 4 (Week 7); T8: Week 12
  Happiness reported assessed objectively by independent observers in session and on videos/photos (0 strongly disagree - 10 strongly agree) using a single-item question (The student feel happy in general).

SECONDARY OUTCOMES:
Change in acculturation | T0: baseline; T2: right before Session 2 (Week 2); T4: right before Session 3 (Week 3); T6: right before Session 4 (Week 7); T8: Week 12
  Three questions about Chinese speaking, interaction with local friends, and watching Chinese Television (TV) programs in the past 7 days (Never, Rarely (1-2 times/week), Occasionally (3-4 times/week), Sometimes (5-6 times/week), Often but not every day (7 times or more/week), Every day: 1-3 times/day, Every day: 4-6 times/day, Every day: 7-9 times/day, Every day: 10 times or more/day).
Change in the ability in speaking Chinese | T0: baseline; T2: right before Session 2 (Week 2); T4: right before Session 3 (Week 3); T6: right before Session 4 (Week 7); T8: Week 12
  A single-item question to ask students their ability in speaking Chinese in the past week (No ability, Simple words or phrases only, A few short sentences, A few short conversations, Some long conversations but not quite fluent, Fluent, Very fluent, Talk like local Chinese).
Change in the attitude in Chinese learning | T1: immediately after Session 1 (Week 1); T3: immediately after Session 2 (Week 2); T5: immediately after Session 3 (Week 3); T7: immediately after Session 4 (Week 7)
  Five questions about the attitude in Chinese and Tang poems. Agreement with the following statements (0 strongly disagree - 10 strongly agree): I like learning Chinese, I am confident in speaking Chinese, I can communicate well in Chinese, I like reciting Tang poems, I am confident in reciting Tang poems.
Parents reported outcomes | T1: immediately after Session 1 (Week 1); T3: immediately after Session 2 (Week 2); T5: immediately after Session 3 (Week 3); T7: immediately after Session 4 (Week 7)
  Three questions about the activity. Do you agree with the following statements (0 Totally Disagree - 10 Totally Agree): Did you enjoy the activity? Do you think your child enjoyed the activity? Do you think your child had fun during the activity?

OTHER OUTCOMES:
Acceptability of the interventions | T1: immediately after Session 1 (Week 1); T3: immediately after Session 2 (Week 2); T5: immediately after Session 3 (Week 3); T7: immediately after Session 4 (Week 7)
  Three questions will asked to the children about their satisfaction (0-10, with "0" indicating "not satisfied at all" and "10" indicating "very satisfied"), willingness to recite Tang poems after the activity and willingness to attend similar activities in the future (0-10, with "0" indicating "no, definitely not" and "10" indicating "yes, definitely yes").
Perceived changes in the attitude in Chinese learning | T1: immediately after Session 1 (Week 1); T3: immediately after Session 2 (Week 2); T5: immediately after Session 3 (Week 3); T7: immediately after Session 4 (Week 7)
  Five questions about their perceived changes after the activity (0 very negative changes - 10 very positive changes) will be asked: interests in learning Chinese, confidence in learning Chinese, fluency in speaking Chinese, interests in reciting Tang poems, and confidence in reciting Tang poems.
Recruitment rate and duration | After recruitment is completed
  The percentage of enrolled participants in the approached participants
Retention rate for each session | T1: immediately after Session 1 (Week 1); T3: immediately after Session 2 (Week 2); T5: immediately after Session 3 (Week 3); T7: immediately after Session 4 (Week 7)
  The percentage of adhered participants in the enrolled participants

CONTACTS AND LOCATIONS:
Overall Officials: Yuying Sun, PhD, Principal Investigator — Hong Kong Metropolitan University
Locations (1):
- Hong Kong Christian Service, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No